CLINICAL TRIAL: NCT02194894
Title: The Effect of Daily Acetaminophen on Patients With Non-alcoholic Fatty Liver Disease (NAFLD) Compared to Healthy Controls
Brief Title: The Effect of Acetaminophen on Non-alcoholic Fatty Liver Disease Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients enrolled
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HS-13-00771
Record Dates: First submitted 2014-06-07; First posted 2014-07-18 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2014-06

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD)
Keywords: Acetaminophen, Non-alcoholic Fatty Liver Disease (NAFLD)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NAFLD patients (Active Comparator): Twenty patients with NAFLD will take 3g of APAP daily for 14 days. Serum liver chemistries and trough acetaminophen (APAP) concentrations will be measured on treatment days 0, 2, 4, 7, 9, 11, 14 and on follow up day 17
  Interventions: Drug: Acetaminophen
- Healthy controls (Active Comparator): Twenty healthy controls will take 3g of APAP daily for 14 days. Serum liver chemistries and trough acetaminophen (APAP) concentrations will be measured on treatment days 0, 2, 4, 7, 9, 11, 14 and on follow up day 17
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — acetaminophen will be given for patient for both arms for 14 days
  Other Names: APAP

SUMMARY:
In this first pilot study, we will examine the effects of acetaminophen dosing in adult patients with NAFLD in comparison to the effects in a healthy control group. Both groups will receive 3 grams (g) of acetaminophen, the maximum recommended daily dose, daily for 14 days. We hypothesize that NAFLD patients are more prone to APAP toxicity than normal controls.Treatment will be stopped after two weeks or in the following conditions:

Treatment with APAP will be stopped in healthy volunteers if ALT and/or AST reached three times the ULN. In patients with NAFLD, treatment will be stopped if: ALT or AST reach ≥ three times the upper limit of entry value or ≥ 5 times the ULN; or if there is ALT or AST >3 times ULN and TBili >2xULN or INR >1.5; or if there is ALT or AST >3 times ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%). We follow a conservative approach derived from the FDA guidelines for stopping medications expected to cause drug induced liver injury (DILI). Indeed, the FDA allows continuation of the medication until ALT or AST are >8x ULN in the absence of elevated Tbili or INR. Patients who have hepatotoxicity will have close monitoring of their liver enzymes until they normalize. Taking acetaminophen up to 3g daily has been shown to be safe and acceptable. We have followed very strict criteria for monitoring and stopping rules however in the usually cases of toxicity the patient will be admitted for monitoring.

ELIGIBILITY:
NAFLD patients:

Inclusion criteria:

1. "Presence of NAFLD": This will be defined by the presence of at least two of the following criteria: (a) suggestion of liver fat by an imaging study (ultrasound, CT scan, MRI or MR spectroscopy) performed in the 6 months prior to enrollment; (b) elevated aminotransferase levels (ALT > 31 U/L for men or > 19 U/L for women, or AST > 30 U/L) on at least two occasions in the 6 months preceding enrollment; and (c) presence of the metabolic syndrome, defined according to the modified AHA/NCEP criteria. Biopsies are not required; however, previous biopsy done within the 6 months prior to the initiation of the study will be considered diagnostic if typical findings of NAFLD are described and other causes of liver disease are ruled out;
2. Individuals who are 18-70 years old;
3. Written informed consent.

Exclusion criteria:

1. Serum ALT > 3 times ULN at baseline.
2. Evidence of another form of liver disease including viral hepatitis, autoimmune hepatitis, cholestatic liver disease, Wilson's disease, Alpha-1-antitrypsin deficiency, hemochromatosis or DILI.
3. History of excess alcohol ingestion, averaging more than 30 gm/day (3 drinks per day) in the previous 10 years, or history of alcohol intake averaging greater than 10 gm/day (1 drink per day: 7 drinks per week) in the previous one year.
4. Evidence of liver cirrhosis on labs or imaging.
5. History of gastrointestinal bypass surgery or ingestion of drugs known to produce hepatic steatosis in the previous 6 months.
6. Significant systemic or major illnesses other than liver disease.
7. Positive test for anti-HIV.
8. Active substance abuse.
9. Pregnancy or inability to practice adequate contraception in women of childbearing potential
10. Evidence of hepatocellular carcinoma.
11. Any other condition which, in the opinion of the investigators, would impede competence or compliance.
12. Serum creatinine >1.5 mg/dl.
13. Starting medications that have been shown to cause drug induced liver injury (eg, augmentin, statins.) within one month prior to enrollment. Medications that have been known to cause DILI but have taken for more than one month prior to enrollment (such as statins) should not be an exclusion.

Healthy Controls:

Inclusion criteria:

1. Individuals who are 18-70 years old
2. Normal Liver enzymes
3. Negative hepatitis B surface antigen, and hepatitis C antibody
4. BMI (18.5 - 24.9) kg/m2
5. Written informed consent.

Exclusion criteria:

1. Presence of the metabolic syndrome, defined according to the modified AHA/NCEP criteria
2. Taking concomitant medications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03-19 (Actual); Study Completion 2015-03-19 (Actual)

PRIMARY OUTCOMES:
This pilot study will seek to answer the question of whether or not NAFLD patients are more prone to APAP toxicity and whether or not lower doses should be recommended. | 14 days
  Liver injury in controls will be defined as an increase in the alanine aminotransferase (ALT) level and/or Aspartae aminotransferase (AST) ≥ three times the upper limit of normal (ULN). Liver Injury in NAFLD patients will be defined as rise of ALT and/or AST ≥3 times baseline levels (which are likely to be elevated) and reaching 5 times ULN. Acetaminophen will be immediately discontinued once the ALT and/or AST reache the defined liver injury level and patients will continue to be monitored. Comparison between the two groups will assess whether or not NAFLD patients are more prone to liver injury than controls.

SECONDARY OUTCOMES:
Exploring possible mechanism of acetaminophen liver injury in NAFLD patients | 14 days
  We plan to measure the serum and urine levels of APAP metabolites including serum levels of acetaminophen-glucuronide (APAP-G) and acetaminophen-sulfate (APAP-S) and the urine levels of cysteine and mercapturic acid conjugates (APAP-C and APAP-M). We also plan to measure APAP protein adducts which are biomarkers of APAP metabolism, reflecting oxidation of APAP and generation of the reactive metabolite NAPQI. We will measure the serum glutathione level and serum markers of mitochondrial injury, including glutamate dehydrogenase (GLDH) and acylcarnitine, as well as markers of necrosis such as miR-122, high-mobility group box-1 protein (HMGB1), full-length keratin 18 and apoptosis marker keratin 18 fragments. The activity of UGT will be estimated by the plasma ratio of APAP-G to APAP at 4 hours (when the first sample is drawn). Expression of CYP2E1 in the peripheral lymphocytes will be assessed using reverse transcription polymerase chain reaction (RT-PCR).

CONTACTS AND LOCATIONS:
Overall Officials: Mazen Noureddin, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - USC, Los Angeles, California
  - USC HCC II (Fatty Liver Clinic), Los Angeles, California